CLINICAL TRIAL: NCT03344107
Title: Comparison Between Symptoms Related to Polaris Loop Stent Versus Vortek Double J Stent After Uncomplicated Flexible Ureterorenoscopy for Renal Stones
Brief Title: Stent-related Symptoms Comparison: Polaris Loop vs Vortek Double-J Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Andrea Bosio, MD Urologist, PhD, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOUCSSTURAB003
Record Dates: First submitted 2017-11-11; First posted 2017-11-17 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Symptoms and Signs; Pain; Renal Calculi
Keywords: Symptoms and Signs; Pain; Renal Calculi; Ureteral Stent; Ureteroscopy
MeSH Terms: conditions — Signs and Symptoms; Pain; Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vortek double-J stent (Active Comparator): Vortek double-J stent after RIRS.
  Interventions: Other: USSQ questionnaire administration after RIRS.
- Polaris Loop stent (Active Comparator): Polaris Loop ureteral stent after RIRS.
  Interventions: Other: USSQ questionnaire administration after RIRS.

INTERVENTIONS:
Other: USSQ questionnaire administration after RIRS. — USSQ symptoms questionnaire administration after RIRS

SUMMARY:
Prospective randomized controlled single-blind parallel-group trial in order to compare symptoms related to loop-tail (Polaris Loop) stents versus conventional double J (Vortek) stents after uncomplicated flexible URS.

DETAILED DESCRIPTION:
Patients undergoing RIRS for a single renal stone < 2 cm are asked to participate in a prospective randomized controlled single-blind parallel-group study. Ureteral stent is always placed after flexible URS. Patients are prospectively randomized into two groups with a 1:1 allocation: group LT receive loop-tail stents (Polaris ™ Loop - Boston Scientific, Natick, USA), while group DJ receive conventional double J stents (Vortek ® - Coloplast, Humlebaek, DK). Stent removal is planned 4 weeks after the procedure.

Participants are asked to fill in the Italian validated version of the Ureteral Stent Symptoms Questionnaire (USSQ) 2 days and 4 weeks after surgery. The USSQ is further submitted 4 weeks after stent removal (8 weeks after surgery) and these results are used as baseline evaluation, on the assumption that SRS persist for a few days after removal.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing flexible ureteroscopy and laser lithotripsy for kidney stones < 2 cm
* given informed consent
* WHO PS 0-2

Exclusion Criteria:

* significant residual fragments at the end of the procedure
* intraoperative complications (i.e. ureteral damage or ureteral stricture)
* urinary tract infections
* anatomic abnormalities
* chronic diseases or medications potentially influencing pain perception and urinary symptoms (i.e. alpha blockers and antimuscarinics)
* preoperative ureteral stenting.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
USSQ Urinary symptoms scores | 4 weeks
  Evaluation of significant differences in Urinary symptoms score between the two groups

SECONDARY OUTCOMES:
USSQ domains scores | 4 weeks
  Evaluation of significant differences in USSQ domains' scores between the two groups
USSQ domains scores | 2 days
  Evaluation of significant differences in USSQ domains' scores between the two groups
USSQ domains' scores adjusted for baseline | 8 weeks
  Evaluation of significant differences in USSQ domains' scores adjusted for baseline between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bosio, MD, Principal Investigator — AOU Città della Salute e della Scienza Torino
Locations (1):
- AOU Città della Salute e della Scienza, Torino, Italy

IPD SHARING:
Plan to Share IPD: No